CLINICAL TRIAL: NCT05453188
Title: Physiotherapy Intervention in Patients With Persistent COVID-19 Disease Using Aerobic Exercise and Association With Genetics
Brief Title: Physiotherapy for Persistent COVID-19 Disease Using Aerobic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URJCLactate
Record Dates: First submitted 2022-07-11; First posted 2022-07-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-07

CONDITIONS: COVID-19; Genetic Predisposition to Disease
Keywords: longCOVID; Aerobic exercise; Muscle performance; Genetics
MeSH Terms: conditions — COVID-19; Genetic Predisposition to Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LongCOVID (Experimental): Patients who have had COVID-19 and have been diagnosed with longCOVID or persistent COVID
  Interventions: Device: Experimental; Genetic: Control
- Control (Active Comparator): Patients who have had COVID-19, but have not been diagnosed with longCOVID or persistent COVID
  Interventions: Device: Experimental; Genetic: Control

INTERVENTIONS:
Device: Experimental — Pre- and post-intervention measurement of quality of life, self-perceived fatigue and blood lactic acid concentration after each Nordic Walking session.
  Other Names: Lactic acid; EuroQool EQ5D; SF-36; MFIS
Genetic: Control — Genetic polymorphism study by Polymerase Chain Reaction (PCR) to determine genetic profile and allele frequencies of patients with persistent COVID and association by Total Genotype Score (TGS) with fatigue status.
  Other Names: ACE polimorphism; ACTN3 polymorphism; AMPD1 polymorphism; CKM polymorphism; MLCK polymorphisms; ACE2 polymorphisms

SUMMARY:
Aerobic exercise - Nordic walking in Persistent Covid (PC) vs. healthy controls.

The main objective of this study is to analyse the genes associated with increased physical performance in patients with PC vs. healthy controls and to measure the level of lactic acid in blood, pre and post exercise session in patients affected by PC.

Relevance: It is intended to be a tool for patients with CP who have not been hospitalised, nor have been offered outpatient rehabilitation treatment. They have not recovered their work, family, sporting or leisure functions. They have particular problems in returning to aerobic exercise.

We think that they may need to be accompanied in the recovery of their physical condition under the supervision of health professionals. Most of the studies offered to them are exploratory, not intervention. Our proposal is a 12-week intervention.

Our proposal, delves into the mechanisms that may underlie their fatigue and their problems in returning to aerobic exercise, in order to collaborate in approaching possible solutions.

Secondary objectives: To study in each of the patients with persistent covid, included in the aerobic Nordic walking programme, their DNA in order to, based on two candidate genes, analyse the role of genetic polymorphisms associated with increased VO2 max training, compared to a healthy control group.

To assess the blood lactic acid level pre and post exercise in a group of patients with persistent covid pre and post aerobic Nordic walking programme. Patients and Methods: 33 patients with CP and 33 healthy controls will follow a Nordic walking programme for 12 weeks. QIAGEN Cube automatic extractor and lactic acid meter will be used.

DETAILED DESCRIPTION:
Design: Parallel non-randomized clinical trial. Study arms: Experimental group with Nordic walking programme (n=15) and healthy control group with the same programme (n=15).

Patients will be recruited by means of a mass mailing to their addresses in the Covid Persistente Madrid group. Participants must meet the inclusion criteria and sign the informed consent form. Patients will be asked to submit a recent basic blood test and an electrocardiogram if available.

Medical Rehabilitation Consultation for screening of patients It is assumed that the patient has already been diagnosed with longCOVID, so he/she should provide data from previous clinical history in relation to the process: time of evolution, characteristics of the syndrome, and treatments carried out.....

It is essential that the patient provides a recent blood test. Objectives To ascertain the main symptomatology presented by the patient, with relevance of signs and symptoms that cause functional limitation.

Determine the presence of comorbidities that may be a contraindication or precaution for the practice of the activity.

The estimated effect size for the main outcome measures established in this project was 0.25. Considering a power of the statistical test of 0.95, an alpha error of 0.05 and a total of five measurements in two participant groups, a minimum number of 30 participants is required, according to the G*Power software (version 3.1.7). Taking into account a loss rate of 10%, the sample size will finally consist of 30 subjects (15 subjects for each intervention group). In order to prevent possible losses, 17 subjects will be included in each group.

5.3. Spatial scope

The assessment will take place:

Consultations with the rehabilitation doctor will take place at the University Clinic of the Faculty of Health Sciences of the Rey Juan Carlos University, Madrid, Spain.

Genetic analysis: Faculty of Health Sciences. Francisco de Vitoria University. Lactic acid measurement: Outdoors, pre- and post-Nordic walking session. Since the measurement must be immediate.

The intervention will take place in the outdoor space of the Casa de Campo. Madrid, Spain.

The Nordic walking sessions will last 90 minutes (warm-up, exercise and cool down), and will be carried out for 12 weeks, with a frequency of once a week.

The instructor will start by designing routes without gradients during the first four sessions of intervention and will adapt the protocol for the following two months according to the evolution of the groups and adapted to the needs of the longCOVID patients.

Patients will be asked to record post-exercise fatigue and their heart rate and oxygen saturation will be monitored during the sessions.

DNA collection for the determination of polymorphisms will be performed on samples to optimize resources (samples will be anonymized and coded).

Samples will be obtained by swabbing and scraping of the buccal mucosa by the participant. DNA will be isolated by QIAGEN Cube automatic extractor. The DNA will be stored at -20º until use.

The genetic study will analyze single nucleotide polymorphisms (SNPs) related fundamentally to functions associated with:

* Polymorphisms of genes associated with muscle performance; ACE, ACTN3, AMPD1, CKM and MLCK
* Polymorphisms of genes for sensitivity and resistance to Covid-19 infection; ACE-2 The data will be entered into the SPSS statistical package (version 25) for analysis.

First, the Kolmogorov-Smirnov test will be used to determine whether the study variables show a normal distribution (p>0.05). Those quantitative variables that do not show a normal distribution will be analysed with non-parametric tests and their data will be expressed as median and interquartile range, while quantitative variables that show a normal distribution will be analysed with parametric tests and their data expressed as mean and standard deviation.

For variables with a normal distribution, a repeated measures analysis of variance (ANOVA) with Bonferroni a posteriori adjustment will be performed, establishing as an inter-subject factor the group parameter (experimental and control) and as an intra-subject factor each of the measurements.

The contrast of variables that do not follow a normal distribution will be carried out using the Mann-Whitney U test, comparing the differences between the groups in each measurement. Intra-group differences will be analysed using the Friedman test for k related samples. In case this test detects intra-group differences at follow-up, the Wilcoxon signed-rank test for two related samples will be used.

Between-group analysis of qualitative variables, expressed as proportions and percentages, will be performed using Pearson's chi-squared test. Intra-group differences of qualitative variables will be performed using McNemar's test for paired data.

The statistical analysis will be carried out with a confidence level of 95%, so that values with a p-value of less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Persistent symptoms of covid for more than one year.
* Age between 30 and 60 years.
* Complete vaccination schedule (one dose is sufficient, as this was considered by the Ministry for patients who have passed the disease).
* Recent basic blood test.

Exclusion Criteria:

* Presence of comorbidities of musculoskeletal origin that contraindicate the practice of the proposed exercise.
* Presence of uncontrolled cardiac or respiratory disease.
* Presence of incapacitating neurological disease that significantly interferes with the proposed exercise activity Severe anaemia or other co-morbidities that significantly interfere with the proposed exercise activity
* Diagnosis or symptoms of dysautonomia
* Presence of high rates of fatigue
* Desaturations during the exercise test that imply a need for oxygen supply for exercise
* Desaturation on exertion during exercise ≥3%.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Lactic acid concentration | Changes from baseline and at the end of procedure (12 weeks)
  A small blood sample (0.3 microlitres) will be taken from the participant, by puncturing the index finger of the hand, to perform a blood lactate analysis. Pre-exercise and immediately after the physical activity
EuroQoL Quality of Life Scale (EQ5D) | Changes from baseline and at the end of procedure (12 weeks)
  The EuroQoL Quality of Life Scale (EQ5D) is an instrument which evaluates the generic quality of life developed in Europe and widely used. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Part II is scored from 0 (worst health state imaginable) to 100 (best health state imaginable). The score from Part II can be used to track changes in health, on an individual or group level, over time
36-Item Short Form Survey (SF-36) | Changes from baseline and at the end of procedure (12 weeks)
  The 36-Item Short Form Survey (SF-36) is a measure of health status and an abbreviated variant of it, the SF-6D, is commonly used in health as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. SF-36 scale is directly transformed into a 0-100 on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Modified Fatigue Impact Scale (MFIS) | Changes from baseline and at the end of procedure (12 weeks)
  The Modified Fatigue Impact Scale (MFIS) is a modified form of the Fatigue Impact Scale based on items derived from interviews with MS patients concerning how fatigue impacts their lives.The total score of the MFIS ranges from 0 to 84. The ranges of scores for each subscale are as follows: physical, 0 to 36; cognitive, 0 to 40; and psychosocial, 0 to 8. A higher score means fatigue is more significantly affecting patient´s life.

SECONDARY OUTCOMES:
Genotype frequency of ACE polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The I/D polymorphism study (rs4340) of angiotensine-converting enzime (ACE) will be used to study blood pressure related to muscle performance.
Genotype frequency of ACTN3 polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The study of the c.1729C>T polymorphism (rs1815739) of alpha-actinine3 (ACTN3) will be used to study the composition of muscle fibres and their relationship with muscle performance.
Genotype frequency of AMPD1 polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The study of the c.34C>T polymorphism (rs17602729) of adenosine monophosphate deaminase 1 (AMPD1) will be used to study muscle metabolism and energy efficiency with its relation to muscle performance.
Genotype frequency of CKM polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The study of the c.*800A>G polymorphism (rs8111989) of muscle-specific creatine kinase (CKM) will be used to study muscle damage during exercise with its relationship to muscle performance.
Genotype frequency of MLCK c.49C>T polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The study of the c.49C>T polymorphism (rs2700352) of myosin-light chain kinase (MLCK) will be used to study muscle damage and loss of strenght during exercise with its relationship to muscle performance.
Genotype frequency of MLCK c.37885C>A polymorphism | Baseline
  Samples shall be obtained by swabbing and scraping of the buccal mucosa by the participant. The study of the c.37885C>A polymorphism (rs28497577) of myosin-light chain kinase (MLCK) will be used to study muscle damage and loss of strenght during exercise with its relationship to muscle performance.
Genotype frequency of ACE2 rs2106806 polymorphism | Baseline
  Samples will be obtained by swabbing and scraping the buccal mucosa by the participant. The study of the angiotensin-converting enzyme 2 (ACE2) rs2106806 polymorphism will be used to study the susceptibility of patients for SARS-CoV-2 infection.
Genotype frequency of ACE2 rs6629110 polymorphism | Baseline
  Samples will be obtained by swabbing and scraping the buccal mucosa by the participant. The study of the angiotensin-converting enzyme 2 (ACE2) rs6629110 polymorphism will be used to study the susceptibility of patients for SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: David Varillas Delgado, PhD, Principal Investigator — Universidad Francisco de Vitoria, crta Pozuelo-Majadahonda km 1.800 PC 28223, Madrid, Spain
Locations (1):
- David Varillas Delgado, Pozuelo de Alarcón, Madrid, Spain